CLINICAL TRIAL: NCT05259202
Title: Value of Fetal Scalp Lactate Sampling During Labour in Cases of Abnormal Fetal Heart Rate During Labor Over 60 Minutes Without a Significant ST-event
Brief Title: Value of Fetal Scalp Lactate Sampling During Labour in Cases of Abnormal Fetal Heart Rate
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL22_0070
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Metabolic Acidosis
Keywords: serious metabolic acidosis; T segment analysis; Blood samples; instrumental delivery; Apgar score; admission to a neonatal ward
MeSH Terms: conditions — Acidosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ST-analysis of the foetal ECG (STAN®) is another second line technique for intrapartum foetal monitoring. Combining ST-analysis with standard CTG interpretation aims to identify hypoxic foetuses more accurately than CTG alone. The STAN® method identifies changes in the ST-interval of the foetal ECG that occur in the presence of foetalcentral hypoxia The aim of this studie is to investigate if the foetal lactate blood sampling is still useful when STAN® monitoring is already being used as a second line technique for intrapartum foetal monitoring if the fetal heart rate is abnormal without a significant ST event Nowadays in the Montpellier hospital's protocol, the investigators have to check the value of lactate sampling in case of le STAN doesn't detect an ST event.

So this studie can change the Montpellier hospital's protocol and avoid useless fetal blood sampling

ELIGIBILITY:
Inclusion criteria:

* patient with labor monitoring by ST segment analysis (STAN) according to current guidelines
* patient who received a fetal lactate sample for fetal heart rate classified as pathological for more than 60 minutes

Exclusion criteria:

* STAN guidelines not respected before installation and during work
* misclassification of fetal heart rate
* obstetrical complications during labor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women monitored by STAN in active labour with singleton term fetus in cephalic presentation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
the incidence of serious metabolic acidosis | day 1
  the incidence of serious metabolic acidosis (defined as pH < 7 and Bdecf > 12 mmol/L in the umbilical cord artery).

SECONDARY OUTCOMES:
Number of the instrumental delivery | day 1
  Apgar score
Number of the neonatal outcome | day 1
  admission to a neonatal ward

CONTACTS AND LOCATIONS:
Overall Officials: WALTZING Aude, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC